CLINICAL TRIAL: NCT05281497
Title: Hemodialysis Health Management Model - the Application of Wearable Devices, Exercise and Nutritional Intervention
Brief Title: Hemodialysis Health Management Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201812145RINA
Record Dates: First submitted 2021-09-26; First posted 2022-03-16 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Physical Inactivity; Nutritional Wasting
Keywords: Hemodialysis; Wearable device; Health management platform
MeSH Terms: conditions — Sedentary Behavior | interventions — Media Exposure; Exercise

STUDY DESIGN:
Intervention Model Description: intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Each participant was provided with a wearable device. Each participant downloaded an app (WowGoHealth app) to connect with the health management platform. All participants were taught to record a dietary diary (taking photos of meals) using a smartphone application. All collected information was uploaded to the health management platform. For the intervention group, we encouraged exercise including an 18-minutes calisthenics. We also built a LINE group to inspire the intervention group.
  Interventions: Behavioral: Health platform; Behavioral: Social media; Other: Exercise training
- Control group (Placebo Comparator): Each participant was provided with a wearable device. Each participant downloaded an app (WowGoHealth app) to connect with the health management platform. All participants were taught to record a dietary diary (taking photos of meals) using a smartphone application. We did not encourage exercise or build a LINE group.
  Interventions: Behavioral: Health platform

INTERVENTIONS:
Behavioral: Health platform — Each participant was provided with a wearable device (a Heart Rate Smart Wristband, GSH405-B6, Golden Smart Home Technology Corporation). Each participant downloaded an app (WowGoHealth app) to connect with the health management platform (GSH AI health platform). Participants' exercise-related data, including number of steps walked, distance, consumed calories, and heart rate, were collected by the wearable devices. All participants were taught to record a dietary diary (taking photos of meals) using a smartphone application. All collected information was uploaded to the health management platform. For the intervention group, we encouraged exercise including an 18-minutes calisthenics made by the Health Promotion Administration, Ministry of Health and Welfare (https://www.youtube.com/watch?v=r3xJW-b2tZY).
Behavioral: Social media — We built a LINE group to inspire the intervention group.
  Arms: Intervention group
Other: Exercise training — exercise including walk and an 18-minutes calisthenics
  Arms: Intervention group

SUMMARY:
Aim: By application of wearable devices and health management platform to strengthen physical activity and improved life quality in hemodialysis patients.

DETAILED DESCRIPTION:
Background: End stage renal disease (ESRD) is a global public health issue. The dialysis therapy brings huge economic burden to many countries. If patients are able to monitor their lifestyle, it not only promotes health, but also reduces the cost of health care.

Aim: By application of wearable devices and health management platform to strengthen physical activity and improved life quality in hemodialysis patients.

Material and Methods: The investigators plan to recruit 30 CKD patients as trial subjects for intervention. The intervention included wearable devices and health management platform for 24 weeks. Patients record their own diet diary by a smartphone application, and their exercise-related data are collected by wearable devices. Then, all the collected information will be upload to health management platform. The investigators compare physical and laboratory examinations before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 20 years and older
* diagnosis of ESRD receiving maintenance HD for more than 3 months

Exclusion Criteria:

* inability to use a smartphone
* impaired walking capacity
* having a psychiatric disorder
* any hospitalization during the previous 3 months.
* has been changing dialysis modality or receiving renal transplantation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change of sit-to-stand-10 (STS-10) | baseline, week 4, week 8, week 12, week 16 and week 24
  time to complete 10 sit-to-stand cycles
Change of sit-to-stand-60 (STS-60) | baseline, week 4, week 8, week 12, week 16 and week 24
  the number of repetitions of sit-to-stand cycles achieved in 60 seconds
Change of 6-minute walking distance (6MWT) | baseline, week 4, week 8, week 12, week 16 and week 24
  the distance the participants walk as fast as they could for 6 minutes on a flat 30-meter track
Change of hand grip strength | baseline, week 4, week 8, week 12, week 16 and week 24
  the strength of hand drip measured by a dynamometer

SECONDARY OUTCOMES:
Change of KDQOL-SF | baseline, week 4, week 8, week 12, week 16 and week 24
  Quality of life measured by the KDQOL-SF (dialysis version)
Change of subjective global assessment (SGA) | baseline, week 4, week 8, week 12, week 16 and week 24
  subjective global assessment for nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yi Li, Study Director — National Taiwan University Hospital
Locations (1):
- Wen-Yi Li, Taipei, Taiwan